CLINICAL TRIAL: NCT03016546
Title: Integrating HIV and Depression Self-Care to Improve Adherence in Perinatal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1204010141; R21MH098667-01A1 (NIH)
Record Dates: First submitted 2017-01-06; First posted 2017-01-10 (Estimated); Last update posted 2020-08-17 (Actual); Status verified 2010-08

CONDITIONS: HIV Infections; Depression
Keywords: Pregnancy
MeSH Terms: conditions — HIV Infections; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BEST-maCARE (Experimental): BEST-maCARE intervention will be refined to accommodate our target population using pertinent information attained through interviews conducted with patients representative of the target group and stakeholders from the clinics where the intervention will be pilot tested.
  Interventions: Behavioral: BEST-maCARE
- time-matched attention control condition (Active Comparator): Participants will be randomly assigned. The control group will receive an intervention that is time and attention equivalent to the experimental condition, though substantively neutral.
  Interventions: Behavioral: Attention Control Condition

INTERVENTIONS:
Behavioral: BEST-maCARE — Features of the integrated BEST-maCARE intervention approach include: Integration of depression screening and linkages to HIV and mental health treatment in the context of perinatal care; A trained, clinic-based nurse (study nurse) plays a mediating role between the health system and its beneficiaries; scheduling of appointments; and, accompanying the patient as needed to initial appointments if desired, and, follow up. Low cost, mobile phone technology is used for frequent one:to:one patient contact with a health care provider (the study nurse) to facilitate continuity of care (for mental health, HIV and pregnancy across the continuum of care from prenatal through postpartum) and promotion of self-care (adherence) and retention in care with a theory-guided, empirically-supported, standardized counseling intervention that is delivered proactively by the study nurse over 18 weeks.
  Arms: BEST-maCARE
Behavioral: Attention Control Condition — The control group will receive an intervention that is time and attention equivalent to the experimental condition. The attention effect that is likely with provision of a mobile phone in the experimental condition will be controlled by providing mobile phone to the control group participants and, they will receive time matched calls from the study nurse with content of the calls focused on infant and maternal nutritional health education per Indian National Guidelines. The phone will be used for delivery of the interventions and may also be used by study staff for purposes of establishing contact or to collect survey interview data if necessary. Time, date, and content of all phone contacts will be documented by the nurse and evaluated in the analysis.
  Arms: time-matched attention control condition

SUMMARY:
Depression is a common perinatal complication that can have a profound, adverse effect on maternal and child health outcomes. The proposed study will directly address this important, but understudied area by evaluating the feasibility and preliminary effect of an innovative, integrated intervention approach, BEST-maCARE [Better Education, Support, Treatment for maternal Capacity, Adherence, REtention in care]. The multi-component intervention is guided by a model drawn from self-regulation and bioecological systems theory. Proactive counseling personalized to the patient and socio-cultural context is delivered by trained clinic personnel (e.g., counselors) to build problem solving and coping skills and linkages to mental health, HIV treatment and ancillary services. The theory-guided intervention approach has been found effective in improving the health behavior and outcomes (e.g., virologic) of vulnerable, marginalized HIV+ women and men in rural and urban settings in the US (AI38858-ACTG 731; R01NR05108). Although the investigators formative research suggests that it is well suited for the target population, its usefulness in addressing significant gaps in care among perinatal women.

l women with co-morbid conditions in a different socio-cultural, limited resource setting has not been studied.

DETAILED DESCRIPTION:
The investigators plan to examine the intervention among perinatal women in Bangalore, India in a two phase developmental study. The theory-guided core elements of the intervention will be maintained, but the content and form of the intervention and study procedures that are context/socio-culturally-specific will be adapted in the first phase of the study to enhance relevance and acceptability among the target population. During the second phase of the project, the investigators will train clinic personnel to deliver the intervention and then pilot test the feasibility, acceptability and fidelity of the novel application of the intervention in a randomized controlled trial. After baseline assessment, participants (n=40) will be randomly assigned to BEST-maCARE or a time-matched attention control condition (each delivered over 18 weeks) and outcomes (e.g., depressive symptoms, adherence) evaluated at 6, 12, 18, and 24 weeks post-randomization.

The specific aims are:

1. Conduct elicitation research with patients and providers in Maharashtra, Delhi, Bangalore and Varanasi, India to gain a more nuanced understanding of the sociocultural context and women's perceived assets and barriers to care to guide adaptation of the Best-maCare intervention protocol to optimize socio-cultural relevance, feasibility and acceptability among perinatal women with co-morbid HIV and depression in this setting.
2. Evaluate the feasibility, acceptability, and fidelity of the study procedures and the adapted, standardized Best-maCare and the attention control conditions and explore their preliminary effect in a randomized, controlled pilot study.

2a) The investigators primary thesis is that the adapted Best-maCare will be feasible and acceptable to women living with HIV in Bangalore, India and other stakeholders. In addition, we expect the fidelity of the intervention will be maintained, and, in keeping with the guiding conceptual framework, that there will be a positive relationship between the Best-maCare intervention and women's medication adherence, engagement in care (HIV, mental health, 6-week postpartum health care services) and health outcomes (HIV-1 RNA, depression, 6-weeks postpartum visit).

The focus of this registration is Aim 2.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant, HIV+ women, in third trimester (≥28 weeks-delivery)
* Eligible for ART treatment or prophylaxis for the PMTCT, during pregnancy, peripartum and postnatal transmission
* screen positive for depressive symptoms
* Speak English, Hindi or Kannada
* Able to provide informed consent.

Exclusion criteria:

* Unable to participate in study visits
* Any condition that, in the opinion of the site investigator, would compromise the candidate's ability to participate.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Program feasibility and acceptability composite | 6 weeks post-delivery
  We will use protocol specific tools to measure feasibility, user acceptability, fidelity and safety of the intervention and study protocol. The assessment will include: 1) The ratio of eligible study participants to those enrolled; 2) Number of scheduled study visits completed; 3) Attrition between baseline and follow-up; 4) Reason for premature drop-out; 5) Number of phone calls that were made on schedule; 6) Level of participation in intervention sessions including the total number sessions, number of sessions completed without break offs, number of break offs, length (minutes) of sessions; 7) Congruence of topic/content discussed on calls with protocol; 8) Patient and study nurse satisfaction with intervention content, mode of delivery, and protocol; 9) Adverse events.
the participant's medication adherence (self-report-ACTG Adherence Questionnaire) | 6 weeks post-delivery
viral load (serum HIV-1 RNA) | 6 weeks post-delivery
depression (self-report-EPDS -Edinburgh Postnatal Depression Scale) | 6 weeks post-delivery
  This scale is a 10-item self-report questionnaire with a possible score range of 0 to 30. Items 1, 2, and 4 are scored 0, 1, 2 or 3 with the top box scored as 0 and the bottom box scored as 3. Items 3 and 5-10 are reverse scored, with the top box scored as 3 and the bottom box scored as 0. The cut-off point for detecting depression was identified as a score of >10. Cases with scores ≥14 were considered to be severely depressed.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Reynolds, Principal Investigator — Yale University School of Nursing
Locations (1):
- Maulana Azad Medical College and Associated Lok Nayak Hospital, G.B. Pant Institute of Postgraduate Medical Education and Research Hospital and Guru Nanak Eye Center, New Delhi, India

IPD SHARING:
Plan to Share IPD: No